CLINICAL TRIAL: NCT06041984
Title: Antiperistaltic Effect and Safety of Glycopyrronium for Colonoscopic Polypectomy: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Antiperistaltic Effect and Safety of Glycopyrronium for Colonoscopic Polypectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jie Chen (Other)
Responsible Party: Sponsor-Investigator, Jie Chen, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023114
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Glycopyrrolate; Colonoscopy
MeSH Terms: interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycopyrrolate (Experimental): Participants will receive intravenous glycopyrrolate 0.2 mg while receiving anesthetic.
  Interventions: Drug: Glycopyrrolate
- Placebo (Placebo Comparator): Participants will receive intravenous 1ml saline while receiving anesthetic.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glycopyrrolate — Intravenous injection of glycopyrrolate 0.2mg
  Arms: Glycopyrrolate
Other: Placebo — Intravenous injection of saline 1ml
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the antiperistaltic effect and safety of glycopyrrolate and whether the use of glycopyrrolate is beneficial for colonoscopy and colonoscopic polypectomy.

DETAILED DESCRIPTION:
Colonic spasm is a major adverse event affecting colonoscopy.The current mainstay for the prevention of colonic spasm is the use of antispasmodic.Glycopyrrolate is a long-acting quaternary ammonium anticholinergic drug.The study is designed as a randomized, double-blind, placebo-controlled study of the efficacy and safety of glycopyrrolate in participants receiving colonoscopy and colonoscopic polypectomy. Patients at our center who met the inclusion criteria were randomized into the glycopyrrolate group and the placebo group, and then statistically analyzed whether there was any difference in the incidence of spasticity, spasticity scores, polyp treatment time, and satisfaction with endoscopist operation between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old.
* Outpatients and inpatients with lesions to be resected under colonoscopy.
* Participants voluntarily participated and signed informed consent forms.

Exclusion Criteria:

* Pregnancy status and lactating women.
* With glaucoma, myasthenia gravis, hyperthyroidism, chronic renal insufficiency, and inflammatory bowel disease.
* With obstructive gastrointestinal diseases such as pyloric obstruction, paralytic ileus, and achalasia of the cardia.
* With obstructive urinary tract diseases such as prostatic hyperplasia and dysuria.
* With heart disease such as arrhythmia (bradycardia, tachycardia, ventricular fibrillation, atrial fibrillation, etc.), coronary heart disease, congestive heart failure.
* With a history of previous abdominal or intestinal surgery.
* Anticholinergic drugs were administered 48 hours before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of intestinal spasm | During Colonoscopy
  The incidence of intestinal spasm in the two groups was calculated after determining whether colonic spasms occurred according to the inhibitory effect score.Rated on a scale of 1 to 3 according to the luminal opening diameter:1 (excellent): no spasm,lumen opening ≥ 2/3 of maximum diameter， 2 (fair): moderate spasm，lumen opening < 2/3 of maximum diameter, but the oral side can be seen and 3 (poor): severe spasm，the oral side lumen is not visible.

SECONDARY OUTCOMES:
inhibitory effect score | During Colonoscopy
  Rated on a scale of 1 to 3 according to the luminal opening diameter:1 (excellent): no spasm,lumen opening ≥ 2/3 of maximum diameter， 2 (fair): moderate spasm，lumen opening < 2/3 of maximum diameter, but the oral side can be seen and 3 (poor): severe spasm，the oral side lumen is not visible.
Polyp Treatment Time | During Colonoscopy
  Time from start of polyp removal to complete polyp removal.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, doctor, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No